CLINICAL TRIAL: NCT00293696
Title: A Randomised Pilot Study to Evaluate the Effect(s) of Casodex 150 mg and Zoladex 3.6 mg on Pathological and Genomic Tumour Markers in Subjects Undergoing Radical Prostatectomy for Localised Prostate Carcinoma
Brief Title: Casodex/Zoladex Biomarkers in Localised Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6876C00001
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Prostate Cancer
Keywords: biomarker study; Patients with clinically localised prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin

INTERVENTIONS:
Drug: bicalutamide (Casodex), goserelin (Zoladex)

SUMMARY:
To evaluate anti-androgen (bicalutamide) induced biological and molecular changes in prostate comparison to chemical castration induced (goserelin) ones

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed localised prostate biopsy specimen that contains sufficient tumour for evaluation of cell proliferation and apoptosis markers
2. Patients who are scheduled for radical prostatectomy with curative intents

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Proliferation by Ki67,
apoptosis marker (TUNEL assay),
Gleason score

SECONDARY OUTCOMES:
expression of known androgen-regulated genes,
biomarkers of apoptotic pathway,
(novel) genomic transcripts

CONTACTS AND LOCATIONS:
Overall Officials: Teuvo L Tammela, Professor, Principal Investigator — Tampere University Hospital
Locations (1):
- TUCH, Tampere, Finland